CLINICAL TRIAL: NCT02646475
Title: Metabolic Effects of Angiotensin-(1-7)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 151699
Record Dates: First submitted 2015-12-31; First posted 2016-01-05 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Insulin Resistance; Hypertension; Metabolic Cardiovascular Syndrome
Keywords: renin-angiotensin system; angiotensin; insulin resistance; blood pressure
MeSH Terms: conditions — Obesity; Insulin Resistance; Hypertension; Metabolic Syndrome | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Angiotensin-(1-7) (Experimental): Subjects will receive intravenous infusion of three ascending doses of Angiotensin-(1-7). The doses are 4, 8, and 16 ng/kg/min. Each dose will be maintained for 10 minutes. The highest dose of Angiotensin-(1-7) will be maintained for an additional 120 minutes during the hyperinsulinemic-euglycemic clamp, for a total of 150 minutes of infusion.
  Interventions: Drug: Angiotensin-(1-7)
- Saline (Placebo Comparator): Subjects will receive an intravenous infusion of saline that is matched in volume to the Angiotensin-(1-7) study day. The saline infusion will also be maintained for a total of 150 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin-(1-7) — This is a biologically active endogenous angiotensin peptide. It may play an important role in the regulation of blood pressure by dilating blood vessels as well as a role in the regulation of insulin action.
  Other Names: Angiotensin I (1-7); Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Normal saline will be used as a placebo comparator.
  Other Names: normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
The overall purpose of this study is to learn more about the metabolic effects of angiotensin-(1-7) in the insulin resistant state associated with obesity. Pharmacologic approaches to increase angiotensin-(1-7) levels or its actions are currently in development for treatment of metabolic-related diseases such as obesity and type II diabetes, based on findings from animal studies. It is unclear if this peptide contributes to the regulation of metabolism in humans. The investigators will test if angiotensin-(1-7) infusion can improve insulin sensitivity measured by hyperinsulinemic-euglycemic clamp methods in individuals with obesity and insulin resistance. The investigators will also examine for changes in blood pressure and related hemodynamic and hormonal changes following angiotensin-(1-7) infusion.

DETAILED DESCRIPTION:
This is an outpatient study that requires a screening visit and two study days in the Vanderbilt Clinical Research Center. Subjects will be asked to stop taking any medications for high blood pressure for at least 2 weeks prior to the study. Subjects will receive intravenous angiotensin-(1-7) or saline infusion on two separate study days, with each study day lasting approximately four hours. There will be at least one week of washout between study days. On each study day, subjects will be instrumented with two intravenous catheters (one for blood sampling and one for drug infusion), arm and finger blood pressure cuffs, and sticky patches to measure heart rate throughout the study. The investigators will take baseline measurements of blood pressure and heart rate and collect blood samples. The investigators will also perform a rebreathing test to measure the heart's pumping capacity. After baseline measurements, the investigators will infuse angiotensin-(1-7) or saline for 30 minutes, with blood pressure and heart rate measured every 10 minutes. At the end of 30 minutes, blood samples will be collected and the rebreathing test will be repeated. The investigators will continue the angiotensin-(1-7) or saline infusion for an additional 2 hours while performing a hyperinsulinemic-euglycemic clamp to measure insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 60 years of age
* Obesity defined as body mass index between 30-40 kg/m2
* Insulin resistance defined as homeostasis model assessment 2 insulin resistance (HOMA2-IR) score >2.2
* Hypertension defined by two or more properly measured seated blood pressure readings >130/85 mmHg, or by use of anti-hypertensive medications. This blood pressure cutoff will allow us to include subjects with pre-hypertension.
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Morbid obesity (BMI > 40 kg/m2)
* Previous allergic reaction to study medications
* Evidence of type I or type II diabetes (i.e. fasting glucose >126 mg/dl, use of anti-diabetic medications)
* Cardiovascular disease other than hypertension such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* History of serious cerebrovascular disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) > 2.0 x upper limit of normal range]
* Impaired renal function (serum creatinine >1.5 mg/dl)
* Anemia (hemoglobin <13.5 g/dl in males or <12.5 g/dl in females)
* Treatment with serotonin-norepinephrine reuptake inhibitors (SNRIs) or norepinephrine transporter (NET) inhibitors
* Treatment with phosphodiesterase 5 inhibitors
* Treatment with anticoagulants
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol (i.e., clinically significant abnormalities on clinical, mental examination or laboratory testing or inability to comply with protocol)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Whole-Body Insulin Sensitivity | steady-state (time 90 to 120 minutes) during hyperinsulinemic-euglycemic clamp
  Whole-body insulin sensitivity will be defined as the glucose infusion rate needed to maintain euglycemia during steady state (time=90 to 120 minutes) of the hyperinsulinemic-euglycemic clamp following angiotensin-(1-7) versus saline infusion. The insulin sensitivity will be corrected by body weight, lean body mass, and steady-state plasma insulin concentrations.

SECONDARY OUTCOMES:
Blood Pressure | 150 minutes
  The change in blood pressure following angiotensin-(1-7) versus saline infusion.
Heart Rate | 150 minutes
  The change in heart rate following angiotensin-(1-7) versus saline infusion.
Cardiac Output | 150 minutes
  The change in cardiac output following angiotensin-(1-7) versus saline infusion.
Stroke Volume | 150 minutes
  The change in stroke volume following angiotensin-(1-7) versus saline infusion.
Systemic Vascular Resistance | 150 minutes
  The change in systemic vascular resistance following angiotensin-(1-7) versus saline infusion.

OTHER OUTCOMES:
Renin Activity | 150 minutes
  The change in plasma renin activity following angiotensin-(1-7) versus saline infusion.
Angiotensin Peptides | 150 minutes
  The change in plasma angiotensin peptides following angiotensin-(1-7) versus saline infusion.
Aldosterone | 150 minutes
  The change in plasma aldosterone following angiotensin-(1-7) versus saline infusion.
Adipokines | 150 minutes
  The change in circulating adipokines following angiotensin-(1-7) versus saline infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Gamboa, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No